CLINICAL TRIAL: NCT07205562
Title: Serum Electrolyte Abnormalities as Prognostic Factor for Outcome in Critically Ill Children
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mennatullah Ahmed Hussein Abdelbary, Principal Investigator, Assiut University
Other Study IDs: Serum Electrolyte Disorders
Record Dates: First submitted 2025-09-17; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Electrolytes Abnormalities; Children; Prognostic Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the clinical profile and outcome of children with serum electrolyte abnormalities admitted at Pediatric Intensive Care Unit in Assuit University Children Hospital.

DETAILED DESCRIPTION:
Electrolyte imbalances are frequent and potentially life-threatening disturbances encountered in pediatric intensive care units (PICUs). These imbalances can reflect underlying pathological processes, treatment interventions, or both, and may influence the clinical course and outcomes of critically ill children. The homeostasis of electrolytes such as sodium, potassium, calcium, and magnesium plays a central role in cellular function, nerve conduction, and cardiovascular stability, making their monitoring and correction crucial during pediatric critical illness .

Studies have highlighted that disturbances like hyponatremia, hyperkalemia, or hypocalcemia often serve as early indicators of disease severity or progression. Kiran and Chaudhary[2021]observed that children admitted with electrolyte abnormalities frequently experienced higher morbidity and mortality compared to those without such disturbances, suggesting a direct correlation with outcomes in the PICU setting .

These abnormalities may arise from diverse etiologies, including dehydration, renal dysfunction, endocrinal disorder and hypothalamic disorder, sepsis, gastrointestinal losses, or medication effects Electrolyte derangements are particularly prevalent among pediatric patients presenting to emergency departments, with age-related differences in presentation and underlying causes. Yen et al. demonstrated that younger children were more prone to sodium and potassium imbalances due to immature renal handling and higher fluid turnover, while older children exhibited abnormalities associated with chronic illnesses or pharmacological agents .Recognizing these patterns can aid in risk stratification and individualized management strategies The spectrum of electrolyte emergencies in children is broad and necessitates rapid identification and intervention. Zieg et al. underscored that life-threatening complications such as arrhythmias, seizures, and cerebral edema often arise from untreated or mismanaged electrolyte disorders, especially in the PICU environment . Hence, early diagnosis and understanding of etiological factors are pivotal in improving clinical outcomes and preventing complications.

Local demographic and regional healthcare factors may also influence the incidence and types of electrolyte abnormalities. In a study from a tertiary care center, Routray et al. found significant variation in electrolyte imbalance profiles across different age groups and disease categories, emphasizing the importance of context-specific evaluation in pediatric populations . Such data are essential for tailoring protocols in resource-limited settings Recent studies such as the one by Rewers et al. on diabetic ketoacidosis have demonstrated that fluid rehydration strategies can impact the rate of correction of acidosis and electrolyte derangements. Their findings highlighted the importance of fluid composition and timing in achieving rapid stabilization without causing further complications . Such protocols are particularly relevant in pediatric patients with metabolic derangements Finally, the overall impact of electrolyte disorders on mortality in the PICU has been underscored in several investigations. Haider et al. found a statistically significant association between electrolyte imbalance and increased risk of death among critically ill children, stressing the need for early intervention and continuous monitoring as part of comprehensive PICU care .

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 month to 18 years.
* Admission to the PICU for any acute medical or surgical reason.
* Availability of serum electrolyte data within the first 24 hours of admission

Exclusion Criteria:

* Children with known chronic kidney disease and chronic liver disease
* Patients with incomplete medical records or missing electrolyte data.
* Children discharged or deceased within 6 hours of admission.
* Patients with chronic liver diseases, or previously diagnosed with adrenal gland disorders

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will include critically ill children admitted to the Pediatric Intensive Care Unit (PICU) at Assiut University Children's Hospital who are found to have serum electrolyte abnormalities during their admission. Patients will be enrolled consecutively over the study period, regardless of gender, aged from 1 month to 18 years.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and Correlation of Electrolyte Abnormalities With PICU Mortality | average of hospital stay: up to 28 days
  To determine the frequency and distribution of electrolyte abnormalities (sodium, potassium, calcium, magnesium, phosphate, and chloride) in critically ill children admitted to the PICU, and to evaluate their correlation with PICU mortality.

SECONDARY OUTCOMES:
Risk Factors and Clinical Outcomes Correlated With Electrolyte Abnormalities in PICU Patients | average hospital stay: up to 28 days
  To identify potentially modifiable risk factors for developing electrolyte abnormalities in critically ill children admitted to the PICU, and to evaluate their correlation with adverse clinical outcomes, including prolonged PICU stay, need for mechanical ventilation, and morbidity indicators (seizures, arrhythmias, altered mental status).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Raza M, Kumar S, Ejaz M, Azim D, Azizullah S, Hussain A. Electrolyte Imbalance in Children With Severe Acute Malnutrition at a Tertiary Care Hospital in Pakistan: A Cross-Sectional Study. Cureus. 2020 Sep 19;12(9):e10541. doi: 10.7759/cureus.10541. PMID 33094080
- [Background] Rewers A, Kuppermann N, Stoner MJ, Garro A, Bennett JE, Quayle KS, Schunk JE, Myers SR, McManemy JK, Nigrovic LE, Trainor JL, Tzimenatos L, Kwok MY, Brown KM, Olsen CS, Casper TC, Ghetti S, Glaser NS; Pediatric Emergency Care Applied Research Network (PECARN) FLUID Study Group. Effects of Fluid Rehydration Strategy on Correction of Acidosis and Electrolyte Abnormalities in Children With Diabetic Ketoacidosis. Diabetes Care. 2021 Sep;44(9):2061-2068. doi: 10.2337/dc20-3113. Epub 2021 Jun 29. PMID 34187840
- [Background] Zieg J, Ghose S, Raina R. Electrolyte disorders related emergencies in children. BMC Nephrol. 2024 Aug 30;25(1):282. doi: 10.1186/s12882-024-03725-5. PMID 39215244
- [Background] Subba Rao SD, Thomas B. Electrolyte abnormalities in children admitted to pediatric intensive care unit. Indian Pediatr. 2000 Dec;37(12):1348-53. No abstract available. PMID 11119337